CLINICAL TRIAL: NCT04059601
Title: Prospective Study on Impact of Preoperative Magnetic Resonance Cholangiopancreatography (MRCP) and Intraoperative Cholangiography (IOC) in Surgical Treatment of Acute Cholecystitis
Brief Title: Magnetic Resonance Cholangiography and Intraoperative Cholangiography in Acute Cholecystitis
Status: Completed | Type: Observational
Sponsor: Jyväskylä Central Hospital (Other)
Responsible Party: Principal Investigator, Olli Helminen, MD, PhD, Jyväskylä Central Hospital
Other Study IDs: Imaging in acute cholecystitis
Record Dates: First submitted 2019-01-03; First posted 2019-08-16 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Acute Cholecystitis
Keywords: common bile duct stones; cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with acute cholecystitis: All patients with acute cholecystitis are included in the study cohort during year 2019. MRCP and IOC will be performed to all patients whenever feasible.
  Interventions: Diagnostic Test: Magnetic resonance cholangiography; Diagnostic Test: Intraoperative cholangiography

INTERVENTIONS:
Diagnostic Test: Magnetic resonance cholangiography — preoperative MRCP in acute cholecystitis before cholecystectomy
Diagnostic Test: Intraoperative cholangiography — Intraoperative cholangiography in acute cholecystitis during cholecystectomy

SUMMARY:
The treatment of choice for acute cholecystitis is cholecystectomy performed as soon as possible after onset of symptoms. Up to 9-22% of patients undergoing cholecystectomy due to cholecystitis have common bile duct stones. Magnetic resonance cholangiopancreatography (MRCP) can aid in technical planning of the operation. Intraoperative cholangiography (IOC) is another method to assess anatomy and stones during operation. There is a lack of quality studies comparing findings of MRCP and IOC and effect on hospital admission.

The aim of this study is to systematically assess the quality of MRCP and IOC in acute cholecystitis, and observe the effect of routine MRCP on surgery outcomes, length of hospital stay, hospital admission costs, and evaluate whether routine IOC could be replaced by MRCP.

DETAILED DESCRIPTION:
Background

The treatment of choice for acute cholecystitis is cholecystectomy performed as soon as possible after onset of symptoms. Early cholecystectomy within 4 days after onset of symptoms resulted in reduced costs, morbidity and shorter hospital stay than delayed cholecystectomy.

Preoperative magnetic resonance cholangiopancreatography ( MRCP) is usually performed if there is a clinical suspicion of common bile duct ( CBD) stones. CBD stones in acute cholecystitis can be found in up to 9-22% of cholecystectomized patients. MRCP in acute cholecystitis can aid in technical planning of laparoscopic cholecystectomy. The benefit of MRCP is the non-invasiveness of the technique with 85-95% sensitivity and 93%-97% specificity.There is a lack of good-quality prospective studies concerning the findings of MRCP and intraoperative cholangiography (IOC) in acute cholecystitis. The purpose of preoperative diagnosis of CBD stones is to facilitate adequate planning of CBD stone removal, which is preferably performed as a single-stage procedure.

In acute cholecystitis the cystic duct may be obliterated and thus cause cannulation difficulties . In these situations preoperative MRCP may give valuable information if CBD stones are present.

The aims of this study is:

1. To observe the feasibility of routine preoperative MRCP in acute cholecystitis in Central Finland Central Hospital
2. To study and compare the quality of MRCP and IOC in acute cholecystitis
3. To study the impact of preoperative MRCP findings in surgical outcome of laparosocpic cholecystectomy

All patients with clinically and radiologically proven acute cholecystitis during one year (2019) will form the study cohort. Ultrasound and MRCP are performed unless there are no contraindications. The quality of MRCP is systematically and independently evaluated by two experienced radiologists. Laparoscopic or open cholecystectomy is programmed and IOC is performed if feasible. The quality and technical success of IOC is recorded and the c-arm cholangiography is documented and stored in the hospital database. In case of common bile duct stones the operating surgeon will decide the policy of stone removal.

The onset of symptoms, hospital arrival, time from arrival to operation, laboratory values, operative details, 30 day morbidity and postoperative outcome are evaluated.

ELIGIBILITY:
Inclusion Criteria:

• Clinically and radiologically confirmed acute cholecystitis

Exclusion Criteria:

* Contraindication for MRCP
* Patients refuses MRCP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in Central Finland Central Hospital district hospitalized and operated due to acute cholecystitis.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
MRCP quality | Hospital admission
  Comparing radiology interobserver findings of preoperative MRCP

SECONDARY OUTCOMES:
Success of intraoperative cholangiography | 1 year
  number of performed intraoperative cholangiographies
preoperative MRCP | 1 year
  proportion of patients with bile duct stones in MRCP
Intraoperative cholangiography | During operation
  Number of patients with bile duct stones in intraoperative cholangiography
Conversion | During operation
  proportion of patients with converted laparoscopic cholecystectomy
Timing of cholecystectomy | hours
  Time gap between onset of symptoms and cholecystectomy
Timing of MRCP | hours
  Time gap between hospital admission and MRCP
Complications | 30 days
  Surgical complications
Length of hospital stay | days
  number of days patients spent in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mattila, MD,PhD, Principal Investigator — Central Finland Central Hospital
Locations (1):
- Central Finland Central Hospital, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Campanile FC, Pisano M, Coccolini F, Catena F, Agresta F, Ansaloni L. Acute cholecystitis: WSES position statement. World J Emerg Surg. 2014 Nov 18;9(1):58. doi: 10.1186/1749-7922-9-58. eCollection 2014. PMID 25422672
- [Result] Roulin D, Saadi A, Di Mare L, Demartines N, Halkic N. Early Versus Delayed Cholecystectomy for Acute Cholecystitis, Are the 72 hours Still the Rule?: A Randomized Trial. Ann Surg. 2016 Nov;264(5):717-722. doi: 10.1097/SLA.0000000000001886. PMID 27741006
- [Result] Blohm M, Osterberg J, Sandblom G, Lundell L, Hedberg M, Enochsson L. The Sooner, the Better? The Importance of Optimal Timing of Cholecystectomy in Acute Cholecystitis: Data from the National Swedish Registry for Gallstone Surgery, GallRiks. J Gastrointest Surg. 2017 Jan;21(1):33-40. doi: 10.1007/s11605-016-3223-y. Epub 2016 Sep 20. PMID 27649704
- [Result] Videhult P, Sandblom G, Rudberg C, Rasmussen IC. Are liver function tests, pancreatitis and cholecystitis predictors of common bile duct stones? Results of a prospective, population-based, cohort study of 1171 patients undergoing cholecystectomy. HPB (Oxford). 2011 Aug;13(8):519-27. doi: 10.1111/j.1477-2574.2011.00317.x. Epub 2011 May 11. PMID 21762294
- [Result] Lee DH, Ahn YJ, Lee HW, Chung JK, Jung IM. Prevalence and characteristics of clinically significant retained common bile duct stones after laparoscopic cholecystectomy for symptomatic cholelithiasis. Ann Surg Treat Res. 2016 Nov;91(5):239-246. doi: 10.4174/astr.2016.91.5.239. Epub 2016 Oct 31. PMID 27847796
- [Result] Tonolini M, Ravelli A, Villa C, Bianco R. Urgent MRI with MR cholangiopancreatography (MRCP) of acute cholecystitis and related complications: diagnostic role and spectrum of imaging findings. Emerg Radiol. 2012 Aug;19(4):341-8. doi: 10.1007/s10140-012-1038-z. Epub 2012 Mar 25. PMID 22447440
- [Result] Romagnuolo J, Bardou M, Rahme E, Joseph L, Reinhold C, Barkun AN. Magnetic resonance cholangiopancreatography: a meta-analysis of test performance in suspected biliary disease. Ann Intern Med. 2003 Oct 7;139(7):547-57. doi: 10.7326/0003-4819-139-7-200310070-00006. PMID 14530225
- [Derived] Mattila A, Helminen O, Pynnonen E, Sironen A, Elomaa E, Nevalainen M. Preoperative MRCP Can Rule Out Choledocholithiasis in Acute Cholecystitis with a High Negative Predictive Value: Prospective Cohort Study with Intraoperative Cholangiography. J Gastrointest Surg. 2023 Nov;27(11):2396-2402. doi: 10.1007/s11605-023-05790-x. Epub 2023 Aug 14. PMID 37578567